CLINICAL TRIAL: NCT04891497
Title: Combination of the Immune Modulator Dimethyl Fumarate With Intraarterial Treatment in Acute Ischemic Stroke
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: There are no suitable patients
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: haojunwei5
Record Dates: First submitted 2021-05-17; First posted 2021-05-18 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2021-05

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Immune Modulator; Dimethyl Fumarate; Intraarterial Treatment
MeSH Terms: conditions — Ischemic Stroke | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraarterial Treatment plus Dimethyl Fumarate (Experimental): Dimethyl fumarate 240mg orally twice daily for 3 consecutive days
  Interventions: Drug: Dimethyl Fumarate
- Intraarterial Treatment plus placebo (Placebo Comparator): Placebo 240mg orally twice daily for 3 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimethyl Fumarate — Dimethyl fumarate 240mg orally twice daily for 3 consecutive days
  Arms: Intraarterial Treatment plus Dimethyl Fumarate
Drug: Placebo — Placebo 240mg orally twice daily for 3 consecutive days
  Arms: Intraarterial Treatment plus placebo

SUMMARY:
The investigators conduct this study to investigate whether oral administration of Dimethyl Fumarate, a Food and Drug Administration-approved drug for multiple sclerosis, is safe and effective in combination with intraarterial treatment in patients with Acute Ischemic Stroke.

ELIGIBILITY:
Inclusion Criteria:

1.18-80 years old 2. NIHSS score>6 3. For the first stroke, MRI showed anterior circulation infarction 4. Patients who meet the mechanical thrombectomy treatment by MRI assessment within 24 hours

Exclusion Criteria:

1. Patients receiving Alteplase thrombolysis
2. Other diseases of the central nervous system
3. There has been a neurological disability in the past (mRS score>2)
4. Difficulty swallowing
5. Arrhythmia, atrioventricular block
6. Use of anti-tumor drugs, other immunosuppressive and immunomodulatory drugs
7. Macular edema
8. Magnetic resonance angiography shows vertebra-basilar artery obstruction
9. Hemorrhagic stroke
10. Patients who are known to have hypersensitivity to dimethyl fumarate or any excipients of this product
11. Pregnant and lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
lesion volume | day 1
  measured by MRI
hemorrhage volume | day 1
  measured by MRI
National Institutes of Health Stroke Scale (NIHSS) | day 1
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.

SECONDARY OUTCOMES:
lesion volume | day3
  measured by MRI
lesion volume | day7
  measured by MRI
lesion volume | day90
  measured by MRI
hemorrhage volume | day3
  measured by MRI
hemorrhage volume | day7
  measured by MRI
hemorrhage volume | day14
  measured by MRI
hemorrhage volume | day90
  measured by MRI
National Institutes of Health Stroke Scale (NIHSS) | day3
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day7
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day14
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
National Institutes of Health Stroke Scale (NIHSS) | day90
  The NIHSS score ranges from 0 to 42 points. The higher the score, the more severe the neurological impairment.
The Modified Rankin Scale (mRS) | day1
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day3
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day7
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day14
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.
The Modified Rankin Scale (mRS) | day90
  The mRS score ranges from 0 to 7 points. The higher the score, the more severe the neurological recovery state of stroke patients.